CLINICAL TRIAL: NCT01055457
Title: Vistakon Investigational Multi-purpose Contact Lens Care Solution.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR-1650
Record Dates: First submitted 2010-01-22; First posted 2010-01-25 (Estimated); Results first posted 2017-01-24 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2017-08

CONDITIONS: Contact Lens Wear

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Experimental Multi-Purpose Solution (Experimental): contact lens care solution
  Interventions: Device: Vistakon Investigational Multi-Purpose Solution II
- ReNu MultiPlus Multi-Purpose Solution (Active Comparator): contact lens care solution
  Interventions: Device: ReNu MultiPlus Multi-Purpose Solution

INTERVENTIONS:
Device: Vistakon Investigational Multi-Purpose Solution II — contact lens care solution
  Arms: Experimental Multi-Purpose Solution
Device: ReNu MultiPlus Multi-Purpose Solution — contact lens care solution
  Arms: ReNu MultiPlus Multi-Purpose Solution

SUMMARY:
This study compares an investigational contact lens care multi-purpose solution to a currently marketed multi-purpose solution.

ELIGIBILITY:
Inclusion Criteria:

* must be an adapted contact lens wearer
* best corrected distance visual acuity must be 20/25 or better in each eye
* must be wearing their habitual lenses on a daily wear basis
* must be willing to refrain from swimming during the study

Exclusion Criteria:

* any systemic diseases that may interfere with contact lens wear
* any clinically significant ocular disease
* any ocular infection
* use of certain medications
* any grade 2 or greater slit lamp findings
* any know sensitivity to marketed contact lens care solutions
* currently pregnant or lactating
* monovision corrected

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2009-11-01 (Actual); Primary Completion 2010-05-01 (Actual); Study Completion 2010-05-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Mission Viejo, California
  - Orlando, Florida
  - Tallahassee, Florida
  - Bloomington, Illinois
  - Pittsburg, Kansas
  - Jamestown, New York
  - Vestal, New York
  - Athens, Ohio
  - Moon Township, Pennsylvania
  - State College, Pennsylvania
  - Amarillo, Texas
  - Katy, Texas
  - Salt Lake City, Utah
  - Charlottesville, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 315 subjects were enrolled in this study. Of the enrolled subjects 20 did not meet the eligibility criteria and 295 subjects were randomized to treatment.Of the randomized subjects 16 were discontinued from the study, while 279 completed the study.
Pre-assignment Details: Allocation of subjects to the 5 contact lenses was fairly balanced ranging from 57 to 61 subjects per lens, while the allocation of subjects to solution was 2:1 for the test and control solution respectively.
Groups:
- Solution1 (Etafilcon A); Solution1 (Comfilcon A); Solution1 (Balafilcon A); Solution1 (Lotrafilcon A); Solution1 (Galyfilcon A): Subjects were random first randomized to 1 of 5 contact lenses and then randomized to receive 1 of 2 contact lens solutions. Solution 1 was an experimental multi-purpose solution.
- Solution2 (Etafilcon A); Solution2 (Comfilcon A); Solution2 (Balafilcon A); Solution2 (Lotrafilcon A); Solution2 (Galyfilcon A): Subjects were random first randomized to 1 of 5 contact lenses and then randomized to receive 1 of 2 contact lens solutions. Solution 2 was ReNu MultiPlus multi-purpose solution.
Period: Overall Study
Arm/Group | Solution1 (Etafilcon A) | Solution1 (Comfilcon A) | Solution1 (Balafilcon A) | Solution1 (Lotrafilcon A) | Solution1 (Galyfilcon A) | Solution2 (Etafilcon A) | Solution2 (Comfilcon A) | Solution2 (Balafilcon A) | Solution2 (Lotrafilcon A) | Solution2 (Galyfilcon A)
Started | 40 | 40 | 38 | 40 | 41 | 18 | 19 | 19 | 20 | 20
Completed | 39 | 39 | 36 | 37 | 38 | 15 | 18 | 18 | 20 | 19
Not Completed | 1 | 1 | 2 | 3 | 3 | 3 | 1 | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 1
Not completed — Subject Disinterest | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Subject Ineligible | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Discomfort | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects that were dispensed a study lens and solution.
Groups:
- Solution 1 (Etafilcon A): All subjects that were dispensed solution 1 and the etafilcon A lens.
- Solution 1 (Comfilcon A): All subjects that were dispensed solution 1 and the comfilcon A study lens.
- Solution 1 (Balafilcon A): All subjects that were dispensed solution 1 and the balafilcon A study lens.
- Solution 1 (Lotrafilcon A): All subjects that were dispensed solution 1 and the lotrafilcon A study lens.
- Solution 1 (Galyfilcon A): All subjects that were dispensed solution 1 and the galyfilcon A study lens.
- Solution 2 (Etafilcon A): All subjects that were dispensed solution 2 and etafilcon A study lens.
- Solution 2 (Comfilcon A): All subjects that were dispensed solution 2 and the comfilcon A study lens.
- Solution 2 (Balafilcon A): All subjects that were dispensed solution 2 and balafilcon A study lens.
- Solution 2 (Lotrafilcon A): All subjects that were dispensed solution 2 and the lotrafilcon A study lens.
- Solution 2 (Galyfilcon A): All subjects that were dispensed solution 2 and the galyfilcon A study lens.
- Total: Total of all reporting groups
Arm/Group | Solution 1 (Etafilcon A) | Solution 1 (Comfilcon A) | Solution 1 (Balafilcon A) | Solution 1 (Lotrafilcon A) | Solution 1 (Galyfilcon A) | Solution 2 (Etafilcon A) | Solution 2 (Comfilcon A) | Solution 2 (Balafilcon A) | Solution 2 (Lotrafilcon A) | Solution 2 (Galyfilcon A) | Total
Number analyzed (Participants) | 40 | 40 | 38 | 40 | 41 | 18 | 19 | 19 | 20 | 20 | 295
Age, Continuous [Mean (Standard Deviation); unit: years]
  Solution 1(etafilcon A) | 30.17 (8.692) | 31.58 (9.459) | 32.16 (8.526) | 29.45 (9.333) | 29.10 (7.993) | 32.48 (7.845) | 29.95 (6.417) | 34.26 (8.738) | 30.10 (9.554) | 32.15 (8.079) | 30.89 (9.012)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 28 | 24 | 25 | 31 | 13 | 9 | 12 | 13 | 9 | 189
  Male | 15 | 12 | 14 | 15 | 10 | 5 | 10 | 7 | 7 | 11 | 106
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 38 | 40 | 41 | 18 | 19 | 19 | 20 | 20 | 295

OUTCOME MEASURES:

1. Primary Outcome: Slit Lamp Findings (SLF)
Description: Slit Lamp Findings were assessed for each subject eye at baseline, 1-day, 1-week, 2-week, 1-month and 3-month follow-up evaluations. SLF consisted of Edema, Corneal Neovascularization, Cornela Staining, Injection, Tarsal Abnormalities and Other findings; each was graded on a 5-likert Scale (Grade: None, Grade 1: Trace, Grade 2: Mild, Grade 3: Moderate and Grade 4: Severe). The number of eyes with Grade 2 or higher across all time points for each SLF variable was reported.
Time Frame: Up to 3 months Post Lens Wear
Population: All subjects that completed the study.
Measure: Number; unit: eyes (2 per subject)
Units Other Than Participants: Subject eyes
Arm/Group | Solution1 (Etafilcon A) | Solution1 (Comfilcon A) | Solution1 (Balafilcon A) | Solution1 (Lotrafilcon A) | Solution1 (Galyfilcon A) | Solution2 (Etafilcon A) | Solution2 (Comfilcon A) | Solution2 (Balafilcon A) | Solution2 (Lotrafilcon A) | Solution2 (Galyfilcon A)
Number analyzed (Participants) | 39 | 39 | 36 | 37 | 38 | 15 | 18 | 18 | 20 | 19
Number analyzed (Subject eyes) | 78 | 78 | 72 | 74 | 76 | 30 | 36 | 36 | 40 | 38
eyes (2 per subject)
  Edema | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Corneal Neovascularization | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Corneal Staining | 8 | 16 | 14 | 12 | 6 | 8 | 3 | 28 | 12 | 8
  Injection | 1 | 0 | 1 | 0 | 3 | 1 | 2 | 4 | 0 | 3
  Tarsal Abnormalities | 15 | 10 | 10 | 10 | 2 | 0 | 1 | 6 | 9 | 1
  Other Findings | 6 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Distance Visual Acuity (LogMAR)
Description: Distance Visual Acuity (LogMAR) was assessed for each subject eye at 1-week, 2-week, 1-month and 3-month follow-up evaluations. The average Visual Acuity (LogMAR) for each time point and lens was reported.
Time Frame: Up to 3 Months Post Lens Wear
Population: All subjects that completed the study.
Measure: Mean (Standard Deviation); unit: LogMAR
Units Other Than Participants: Subjects Eyes
Arm/Group | Solution1 (Etafilcon A) | Solution1 (Comfilcon A) | Solution1 (Balafilcon A) | Solution1 (Lotrafilcon A) | Solution1 (Galyfilcon A) | Solution2 (Etafilcon A) | Solution2 (Comfilcon A) | Solution2 (Balafilcon A) | Solution2 (Lotrafilcon A) | Solution2 (Galyfilcon A)
Number analyzed (Participants) | 39 | 39 | 36 | 37 | 38 | 15 | 18 | 18 | 20 | 19
Number analyzed (Subjects Eyes) | 78 | 78 | 72 | 74 | 76 | 30 | 36 | 36 | 40 | 38
LogMAR
  1-week | -0.033 (0.0601) | -0.042 (0.0630) | -0.037 (0.0563) | -0.040 (0.0665) | -0.029 (0.0615) | -0.055 (0.0580) | -0.033 (0.0601) | -0.040 (0.0540) | -0.045 (0.0685) | -0.012 (0.0619)
  2-week | -0.045 (0.0642) | -0.041 (0.0663) | -0.047 (0.0592) | -0.039 (0.0649) | -0.037 (0.0594) | -0.058 (0.0585) | -0.045 (0.0642) | -0.051 (0.0625) | -0.031 (0.0551) | -0.030 (0.0595)
  1-Month | -0.045 (0.0623) | -0.042 (0.0644) | -0.033 (0.0658) | -0.040 (0.0628) | -0.037 (0.0595) | -0.068 (0.0541) | -0.045 (0.0623) | -0.026 (0.0534) | -0.031 (0.0626) | -0.032 (0.0610)
  3-Month | -0.045 (0.0673) | -0.031 (0.0609) | -0.039 (0.0617) | -0.038 (0.0607) | -0.031 (0.0613) | -0.051 (0.0668) | -0.045 (0.0673) | -0.034 (0.0567) | -0.014 (0.0618) | -0.040 (0.0614)

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study. Approximately 3 months.
Arm/Group | Solution1 (Etafilcon A) | Solution1 (Comfilcon A) | Solution1 (Balafilcon A) | Solution1 (Lotrafilcon A) | Solution1 (Galyfilcon A) | Solution2 (Etafilcon A) | Solution2 (Comfilcon A) | Solution2 (Balafilcon A) | Solution2 (Lotrafilcon A) | Solution2 (Galyfilcon A)
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/38 | 1/40 | 0/41 | 0/18 | 0/19 | 0/19 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/38 | 0/40 | 2/41 | 0/18 | 1/19 | 1/19 | 0/20 | 1/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Solution1 (Etafilcon A) (N=40) | Solution1 (Comfilcon A) (N=40) | Solution1 (Balafilcon A) (N=38) | Solution1 (Lotrafilcon A) (N=40) | Solution1 (Galyfilcon A) (N=41) | Solution2 (Etafilcon A) (N=18) | Solution2 (Comfilcon A) (N=19) | Solution2 (Balafilcon A) (N=19) | Solution2 (Lotrafilcon A) (N=20) | Solution2 (Galyfilcon A) (N=20)
Vitreous Hemorrhage / Retinal Detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Solution1 (Etafilcon A) (N=40) | Solution1 (Comfilcon A) (N=40) | Solution1 (Balafilcon A) (N=38) | Solution1 (Lotrafilcon A) (N=40) | Solution1 (Galyfilcon A) (N=41) | Solution2 (Etafilcon A) (N=18) | Solution2 (Comfilcon A) (N=19) | Solution2 (Balafilcon A) (N=19) | Solution2 (Lotrafilcon A) (N=20) | Solution2 (Galyfilcon A) (N=20)
Conjunctivitis - Bacterial (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Symptoms/ Complaints (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) — Symptoms and complaints requiring treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days